CLINICAL TRIAL: NCT01611220
Title: Dissonance Inpatient Relapse Prevention Program for Anorexia Nervosa: A Randomized Control Trial
Brief Title: Dissonance Inpatient Relapse Prevention Program for Anorexia Nervosa
Acronym: RePAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Garda Hospital (Other)
Responsible Party: Principal Investigator, Riccardo Dalle Grave, Head of Department of Eating and Weight Disorders, Villa Garda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USL22#03/12-CEP329
Record Dates: First submitted 2012-05-25; First posted 2012-06-04 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Relapse prevention; Cognitive Dissonance; Inpatient treatment; Cognitive behavior therapy
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard cognitive behavior inpatient treatment
- RePAN (Experimental): Standard cognitive behavior inpatient treatment plus 8 dissonance relapse prevention groups
  Interventions: Behavioral: RePAN

INTERVENTIONS:
Behavioral: RePAN — The dissonance relapse prevention intervention consists of eight groups conducted by a psychologist who involves participants in interactive activities aimed to prevent relapse after discharge from the inpatient treatment
  Other Names: Dissonance relapse prevention
  Arms: RePAN

SUMMARY:
Anorexia Nervosa inpatient treatment has often a short-term success as weight is restored to a healthy level, but high percentage of patients relapse during the first year following the discharge. The development of strategies to overcome this problem represents a priority for clinicians. Aim of this trial is to evaluate the effects of a relapse prevention program based on cognitive dissonance theory developed for hospitalized patients.

DETAILED DESCRIPTION:
Inpatient treatment for anorexia nervosa is often successful in restoring body weight, but a high percentage of patients relapse following discharge. The aim of the study was to assess the effect of a relapse prevention program during the last phase of inpatient treatment. Patients, when they achieve a BMI of 18.5, are randomly allocated to complete the standard cognitive behavior inpatient treatment (CBT-I) or to complete the standard CBT-I plus eight relapse prevention groups based on the cognitive dissonance. The intervention has been derived by the selective and indicated prevention programs using a dissonance-based approach. This intervention showed to be effective in reducing the risk for eating pathology onset. The primary outcome of the study is to assess the number of patients allocated to the two condition with a BMI equal or greater than 18.5 at 12-months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Body Mass Index ≥ 18.5
* Anorexia Nervosa patients admitted to inpatient treatment
* Written informed consent

Exclusion Criteria:

* Male
* Schizophrenia or other psychiatric disorders
* Substance abuse
* Medical complication that may hamper the interpretation of results (medical condition that causes weight changes)
* Absence of medical treatment (drugs) that may hamper the interpretation of results
* Pregnancy or plan to get pregnant

Ages: 13 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 1 year
  The main outcome is to assess the number of patients with good BMI outcome (BMI ≥ 18.5) at 12-month follow-up end in the two arm conditions.

SECONDARY OUTCOMES:
Eating disorder Examination (EDE) | 1 year
  Number of patients with "full remission" defined as having a global EDE score below 1SD above the community mean (1.74) and a BMI ≥ 18.5.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Dalle Grave, MD, Principal Investigator — Department of Eating and Weight Disorders, Villa Garda Hospital
Locations (1):
- Villa Garda Hospital, Garda, Verona, Italy

REFERENCES:
- [Background] Stice E, Marti CN, Spoor S, Presnell K, Shaw H. Dissonance and healthy weight eating disorder prevention programs: long-term effects from a randomized efficacy trial. J Consult Clin Psychol. 2008 Apr;76(2):329-40. doi: 10.1037/0022-006X.76.2.329. PMID 18377128